CLINICAL TRIAL: NCT02208427
Title: Toward a Safe and Reachable Preventive Therapy for LTBI: a Multicenter Randomized Controlled Study in Taiwan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201309055MINC
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Latent Tuberculosis Infection
Keywords: isoniazid, LTBI, rifapentine, TST
MeSH Terms: conditions — Latent Tuberculosis | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3M_RH (Experimental): Rifapentine and Isoniazid for 3 months: weekly oral rifapentine 15 mg/kg plus isoniazid 15 mg/kg for 12 doses
  Interventions: Drug: Rifapentine and Isoniazid for 3 months
- 9M_INH (Active Comparator): Isoniazid for 9 months: daily oral isoniazid 5 mg/kg for 9 months
  Interventions: Drug: Isoniazid for 9 months

INTERVENTIONS:
Drug: Rifapentine and Isoniazid for 3 months — weekly oral Rifapentine 15 mg/kg plus Isoniazid 15 mg/kg for 12 doses
  Other Names: Priftin; Isoniazid
  Arms: 3M_RH
Drug: Isoniazid for 9 months — daily oral Isoniazid 5 mg/kg for 9 months under supervision (conventional IPT)
  Other Names: Isoniazid
  Arms: 9M_INH

SUMMARY:
Background:

Tuberculosis (TB) remains the most important infectious disease in the world. Keys to successful control of TB is rapid diagnosis, prompt treatment, as well as effective preventive therapy for contacts with latent TB infection (LTBI). Current methods for the diagnosis of LTBI are tuberculin skin test (TST) and interferon-gamma release assay (IGRA). For preventive therapy, the recommended regimens include daily isoniazid for 9 months and daily rifampicin for 4 months. By incorporating long-acting rifapentine, a new regimen combining weekly rifapentine and high-dose isoniazid for a total of 12 doses has been proven of equal potency and toxicity. However, the treatment completion rate is much higher in weekly treatment for 3 months than daily treatment for 9 months. It is reasonable that using rifapentine-based preventive therapy can markedly increase the completion rate. However, study is lacking, especially in Asia, the high endemic area of TB.

With the effort of all health care workers and public health personnel, the incidence of TB in Taiwan has gradually declined in recent 10 years. In order to maintain the trend of decreasing in incidence, preventive therapy for LTBI become more and more important. However, which is the best preventive regimen for LTBI is still unknown. Therefore, we conduct the prospective randomized multicenter studies to compare the treatment completion rate of two regimens in Taiwan. The first regimen is daily isoniazid for 9 months. The second is weekly rifapentine plus high-dose isoniazid for 3 months.

DETAILED DESCRIPTION:
Background:

Tuberculosis (TB) remains the most important infectious disease in the world. Keys to successful control of TB is rapid diagnosis, prompt treatment, as well as effective preventive therapy for contacts with latent TB infection (LTBI). Current methods for the diagnosis of LTBI are tuberculin skin test (TST) and interferon-gamma release assay (IGRA). For preventive therapy, the recommended regimens include daily isoniazid for 9 months and daily rifampicin for 4 months. By incorporating long-acting rifapentine, a new regimen combining weekly rifapentine and high-dose isoniazid for a total of 12 doses has been proven of equal potency and toxicity. However, the treatment completion rate is much higher in weekly treatment for 3 months than daily treatment for 9 months. It is reasonable that using rifapentine-based preventive therapy can markedly increase the completion rate. However, study is lacking, especially in Asia, the high endemic area of TB.

With the effort of all health care workers and public health personnel, the incidence of TB in Taiwan has gradually declined in recent 10 years. In order to maintain the trend of decreasing in incidence, preventive therapy for LTBI become more and more important. However, which is the best preventive regimen for LTBI is still unknown. Therefore, we conduct the prospective randomized multicenter studies to compare the treatment completion rate of two regimens in Taiwan. The first regimen is daily isoniazid for 9 months. The second is weekly rifapentine plus high-dose isoniazid for 3 months.

Specific Aims:

1. Understanding which of the two preventive regimens has the highest completion rate under supervision.
2. Understanding the reasons of interruption in preventive therapy.
3. Comparing the side effect profile of the two preventive regimens in Taiwan.

Methods:

In this prospective multicenter study, we will enroll close contacts aged >=12 with positive TST. Chest radiography and sputum studies, if necessary, will be performed to exclude active pulmonary TB. After performing baseline IGRA, participants will be randomized into 2 groups with different preventive regimens. The first regimen is daily isoniazid for 9 months. The second is weekly rifapentine plus high-dose isoniazid for 3 months. The primary outcome is treatment completion rate of the two preventive regimens. The secondary outcome is toxicity. All participant will be followed for 2 years and screen for the development of active pulmonary TB by chest radiography and sputum studies if necessary. The reasons for treatment incompletion will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Household contacts of TB or TB contacts in schools or densely-populated institutes
* Age ≥12 year-old
* Index case having smear-positive pulmonary TB
* Contact with index case for >8 hours within single day or >40 hours within total transmissible period
* TST ≥10 mm within one month
* Born in 1986 or after (not applicable in the National Taiwan University Hospital Hsin-Chu branch and Chang-Hua Hospital)

Exclusion Criteria:

* Clinical or radiographic evidence of active TB
* Index case having culture-negative pulmonary TB
* Index case having Isoniazid or Rifampin-resistant TB
* Receiving medications with significant interactions with Isoniazid, Rifampin, or Rifapentine
* Allergy to Isoniazid, Rifampin, or Rifapentine
* Sero-positive for hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Documented liver cirrhosis
* Human immunodeficiency virus (HIV) infection
* Receiving immunosuppressants
* Receiving biological agents
* Hemoglobin <8 g/dL
* Neutrophil <750000 /mL
* Total bilirubin >2.5 mg/dL
* Aspartic transaminase (AST) or alanine transaminase (ALT) >2 folds of upper limit of normal (ULN)
* Pregnant or breast-feeding
* Life expectancy <3 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
completion rate | 2 years
  This prospective randomized interventional study is aimed to assess the completion rate of two different preventive regimens for LTBI by intent-to-treat analysis. Interruption of preventive therapy due to any reasons will be considered as incompletion.

SECONDARY OUTCOMES:
side effect | 3 months in the 3M_RH group and 9 months in the 9M_INH group
  To evaluate the side effect profile (especially hepatotoxicity, defined as AST and/or ALT ≥2 ULN) of the two preventive regimens
interruption | 3 months in the 3M_RH group and 9 months in the 9M_INH group
  To calculate the number of participants with interruption in preventive therapy and to know the reasons of interruption by questionnaire
active TB | 2 years after enrollment
  To know the rate of active TB within subsequent 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, MD. PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun HY, Huang YW, Huang WC, Chang LY, Chan PC, Chuang YC, Ruan SY, Wang JY, Wang JT. Twelve-dose weekly rifapentine plus isoniazid for latent tuberculosis infection: A multicentre randomised controlled trial in Taiwan. Tuberculosis (Edinb). 2018 Jul;111:121-126. doi: 10.1016/j.tube.2018.05.013. Epub 2018 Jun 7. PMID 30029896